CLINICAL TRIAL: NCT03064659
Title: Driving Pressure And Limitation of Expiratory Flow: Evaluation of Postoperative Pulmonary Complications in Elective Adult Cardiac Surgery.
Brief Title: Driving Pressure And EFL in Adult Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Elena Bignami, MD, Ospedale San Raffaele
Other Study IDs: DPEFLCCH
Record Dates: First submitted 2017-02-17; First posted 2017-02-27 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure; Pneumothorax; Atelectasis; Respiratory Infection; Bronchospasm; Pleural Effusion
Keywords: Postoperative pulmonary complications; Driving Pressure; Limitation of Expiratory Flow; Cardiac Surgery; Cardio-pulmonary bypass
MeSH Terms: conditions — Respiratory Insufficiency; Pneumothorax; Pulmonary Atelectasis; Respiratory Tract Infections; Bronchial Spasm; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During general anesthesia, functional residual capacity (FRC) is reduced. If the FRC is lower than the minimum volume required to maintain the opening of the airways, there is a derecruitment of the lung parenchyma, leading to the phenomenon of expiratory flow limitation (EFL).

The Driving Pressure (DP) is the difference between the plateau pressure (Pplateau) and the Positive End-Expiratory Pressure (PEEP), and estimates the lung strain.

The incidence of EFL and the importance of DP are not known in adult cardiac surgery, so it's necessary a study to assess both. The primary end-point of the study is to evaluate the correlation of DP and EFL with PPCs in adult cardiac surgery. The secondary end-point of the study is to evaluate: the mechanical ventilation time, the length of ICU and hospital stay, the rehospitalization and mortality.

It will be a prospective, observational, non-pharmacological study. It will enroll 200 patients undergoing elective adult cardiac surgery.

DETAILED DESCRIPTION:
During general anesthesia, functional residual capacity (FRC) is reduced. If the FRC is lower than the minimum volume required to maintain the opening of the airways (closing capacity), there is a derecruitment of the lung parenchyma, leading to the phenomenon of expiratory flow limitation (EFL). Numerous factors contribute to the EFL, including hyperoxia, muscle paralysis, the increase of the volume of the interstitial fluids and the inflammatory response.

To establish the presence of EFL under general anesthesia, it was developed a test known as PEEP test. It is the sudden removal of 3 cm H2O to the value of positive end-expiratory pressure (PEEP test): in the EFL the subtraction of the expiratory pressure does not produce an increase of expiratory flow. The use of different modality of mechanical ventilation during cardiac surgery may impact on the incidence of EFL post CEC.

The Driving Pressure (DP) is the difference between the plateau pressure (Pplateau) and the Positive End-Expiratory Pressure (PEEP), and estimates the lung strain.

The primary end-point of the study will be:

- Evaluate the correlation of DP and EFL with PPCs in patients undergoing elective cardiac surgery performed with extracorporeal circulation.

The secondary end-point of the study will be:

* Consider whether there are factors associated with the development of EFL, especially comorbidities and ventilation mode during surgery;
* Evaluate outcomes such as duration of mechanical ventilation, length of stay in intensive care (ICU), PaO2/ FiO2 at discharge from the ICU, development of respiratory complications, duration of hospital stay and mortality.

It will be a prospective, observational, non-pharmacological study. It will enroll 200 patients undergoing elective adult cardiac surgery.

Respiratory rate will be set to maintain PaCO2 at values close to eucapnia. It will be used to pressure-controlled ventilation (Pinsp ≤ 35 cm H2O) only if the controlled ventilation is reached and exceed the maximum airway pressures. In this case it will be necessary to check that the volume delivered by the ventilator is really, for the entire period, the chosen volume. The inspiratory way will be composed of O2, air and maybe the halogenated anesthetic. The O2 concentration will be increased gradually in case of desaturation up to maintain SpO2 93-95% trying not to exceed the FiO2 of 0.8 if it will be choice a protective ventilation strategy.

Weaning from the CEC will include a single alveolar recruitment maneuver, in which the airway pressure will be increased to 40 cm H20 for 7 seconds.

At the end the patients will be transferred to the Intensive Care Unit (ICU) for post-operative monitoring. During the transfer will be supported with mechanical ventilation performed manually by the anesthetist resuscitator.

Extubation in ICU will run in according to the protocol of the center. It could be used any postoperative analgesia that provides NRS at rest ≤ 3 and dynamic NRS (cough) ≤ 4 and allow an active chest physical therapy (CPT).

The following information will be collected:

In the section devoted to the preoperative treats will be fit the patient data related to:

* Age, weight, height, sex;
* Comorbidities
* Positive respiratory history of: previous pleural-parenchymal disease within 30 days prior to the intervention, previous surgery of the thorax, pleura or lung, presence of pleural effusion;
* History of smoking cigarettes: Active smoking (number of cigarettes), ex-smoker or non-smoker;
* SpO2, PaO 2, PaO 2 / FiO 2, PaCo 2 (if available);
* Cardiological history (echocardiography, ECG, etc.)
* Other medical history information of relevance to the study

In the dedicated intraoperatory tab will be collected the following data:

* Incidence of EFL and respiratory mechanics parameters;
* Type of surgery;
* Time to CEC, clamping, cardioplegia, type of circuit and oxygenator;
* Transfusion of blood products;
* Any administration of cardio / vasoactive drugs;
* Duration of surgery;
* Other information relevant for the purposes of the study.

In the schedule about the post-operative treats will be collected the following data:

* Postoperative mechanical ventilation time;
* Postoperative respiratory complications;
* Postoperative non-respiratory complications (cardiovascular, infectious, kidney, surgical);
* The need for re-intubation in the postoperative period;
* The need for ventilatory support (non-invasive ventilation, invasive ventilation) in the postoperative period;
* Need for hospitalization in intensive care (expected, unexpected, cause of hospitalization, length of stay);
* Length of hospital stay;
* Other information about the postoperative relevant to the study The study does not interfere with the normal anesthetic activity, it does not provide for variations from the procedures currently used and the PEEP test use does not involve pathophysiological changes for the patient.

Data will be collected on the appropriate Case Report Form (CRF). It will be collected anamnestic information, data about surgery and post-operative clinical data, in particular respiratory parameters. Definitions and use of outcome measures are in according to the standards for European Perioperative Clinical Outcome (EPCO) definitions [Eur J Anaesthesiol 2015; 32:88-105].

Data will be analyzed with a professional statistical software. Univariate and multivariate analysis will be performed. Chi-square test will be used for dichotomous variables, z-test/t-test or the Mann-Whitney U-test for continuous variables, as appropriate. Statistical significance if p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Ability to provide an informed consent
* Planned cardiac surgery with median sternotomy and bi-pulmonary ventilation
* patients scheduled for adult elective cardiac surgery, performed with CPB and aortic cross-clamping.

Exclusion Criteria:

* Patient refusal to provide informed consent
* Emergency surgery
* Cardiac surgery with TAVI/MitraClip
* Planned thoracotomy with one lung ventilation
* Patients with chronic kidney insufficiency (defined as dialysis)
* Patients already intubated in the peri-operative period
* Patients with pneumonia in the pre-operative period (30 days before surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Undergoing Elective Cardiac Surgery
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Expiratory Flow Limitation | Through study completion, an average of 24 hours after surgery
Incidence of Driving Pressure | Through study completion, an average of 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative pulmonary complication | Through study completion, an average of 7 days after surgery
  Respiratory Failure, Pneumothorax, Atelectasis, Respiratory Infection, Bronchospasm, Pleural Effusion
ICU length of stay | Through study completion, an average of 24 hours after surgery
Hospital length of stay | Through study completion, an average of 7 days after surgery
Duration of mechanical ventilation | Through study completion, an average of 7 days after surgery
PaO2/ FiO2 | Through study completion, an average of 24 hours after surgery
Mortality | Through study completion, an average of 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elena Bignami, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

REFERENCES:
- [Background] Grieco DL, Chen L, Dres M, Brochard L. Should we use driving pressure to set tidal volume? Curr Opin Crit Care. 2017 Feb;23(1):38-44. doi: 10.1097/MCC.0000000000000377. PMID 27875410